CLINICAL TRIAL: NCT04908137
Title: Use of 2-Octyl Cyanoacrylate (Dermabond) in Neonatal Circumcision: A Randomized Controlled Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Michael Chua, Staff Urologist, The Hospital for Sick Children
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1000070281
Record Dates: First submitted 2021-05-26; First posted 2021-06-01 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Redundant Prepuce
Keywords: Circumcision
MeSH Terms: interventions — octyl 2-cyanoacrylate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2-Octyl Cyanoacrylate (Dermabond) Group (Experimental): 2-Octyl Cyanoacrylate (Dermabond) 0.5ml/ sticks topical application around post-circumcision site subcoronal area immediately after the circumcision devise is removed and circumcision procedure was done
  Interventions: Drug: 2-octyl cyanoacrylate
- Control Group (No Intervention): will receive Vaseline cream application around the post-circumcision site immediately after circumcision

INTERVENTIONS:
Drug: 2-octyl cyanoacrylate — Topical Skin Adhesive is a sterile, liquid topical skin adhesive containing a monomeric (2-octyl cyanoacrylate) formulation and the colorant D & C Violet No. 2. It is provided as a single use applicator in a blister package
  Other Names: Dermabond
  Arms: 2-Octyl Cyanoacrylate (Dermabond) Group

SUMMARY:
Study Description: 2-Octyl Cyanoacrylate (Dermabond) use in neonatal circumcision are being practiced to prevent complications; however, no randomized controlled trials was ever done to assess efficacy and safety. This is a single-centered, randomized clinical trial to assess the efficacy and safety of 2-Octyl Cyanoacrylate (Dermabond) application in neonatal circumcision to prevent complication.

Primary Objective: To determine the efficacy and safety of 2-Octyl Cyanoacrylate (Dermabond) application versus control in neonatal circumcision to prevent post-procedural complication.

Secondary Objectives:

1. To assess post-procedural pain score difference between with versus without 2-Octyl Cyanoacrylate (Dermabond) application in neonatal circumcision
2. To assess parents' satisfaction and cosmesis post-neonatal circumcision with versus without 2-Octyl Cyanoacrylate (Dermabond) application.

Endpoints: Primary Endpoint: Complication rates post-neonatal circumcision within 180 days with the following complication in specific or in composite ⦁ Bleeding requiring hemostatic intervention (suturing, dermabond application, silver nitrite application, pressure bandage)

* Infection requiring antibiotic administration or wound drainage
* Excess skin as assessed by parents satisfaction
* Meatal stenosis
* Adhesion requiring surgical correction.

Secondary Endpoints:

1. pain score within 5 min and 30 minutes postneonatal circumcision using the FLACC score by parents and MBPS scale by a medical allied personnel.
2. Parents satisfaction as determined by a simple 10-score liked scale and cosmesis assessment scale within 24hrs and within 30 days post-neonatal circumcision. Complication rates detailed above in specific time points clustered according to (within 24 hrs, within 2 weeks, within 30 days, within 30 to 180 days).

Study Population: 280 male neonates (140 each intervention groups) who are eligible for neonatal circumcision with no other medical co-morbidities.

Intervention:

2-Octyl Cyanoacrylate (Dermabond) 0.5ml/ sticks) topical application around post-circumcision site subcoronal area.

ELIGIBILITY:
Inclusion Criteria:

* Consent provided by one of the parents
* Male sex eligible for neonatal circumcision (with no genital anomalies, such as hypospadias components or congenital curvatures)
* Aged 2 to 60 days
* In good general health as evidenced by medical history
* No history of hematological diseases with clotting or bleeding disorders such as hemophilia, Von Willebrand diseases

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Presence of bleeding or clotting disorders
  * Family history of bleeding or clotting disorder
  * Genital anomalies such as hypospadias, severe ventral curvatures
  * Known allergic reactions to components of the 2-Octyl Cyanoacrylate (Dermabond)
  * Febrile illness within 48hrs
  * Any condition or diagnosis, that could in the opinion of the Principal Investigator or the delegate interfere with the participant's ability to comply with study instructions, might confound the interpretation of the study results, or put the participant at risk.

Ages: 2 Days to 60 Days | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 280 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Complication rates (Composite) | 180 days post neonatal circumcision
  Composite complication rates post-neonatal circumcision within 180 days following neonatal circumcision

SECONDARY OUTCOMES:
Pain score (FLACC) by Parents | 5 minutes and 30 minutes
  pain score within 5 minutes post-neonatal circumcision using the FLACC score by parents. (Higher Score is Worse)
Pain score (MBPS) by Medical Personnel | 5 minutes and 30 minutes
  pain score within 5 minutes and 30 minutes post-neonatal circumcision using the MBPS scale by a medical allied personnel. (Higher Score is Worse)
Parents Satisfaction | within 24 hours and 30 days post neonatal circumcision
  Parents satisfaction as determined by a simple 10-score liked scale and cosmetic assessment scale within 24hours and within 30 days post-neonatal circumcision
Complication rates (specific case characteristics) | within 24 hours, within 2 weeks, within 30 days within 30 to 180 days
  Complication rates post-neonatal circumcision

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No